CLINICAL TRIAL: NCT06653829
Title: NST-SPARK: Preliminary Study of an Augmented Reality (AR) App Delivering Recovery-Oriented Cognitive Therapy for Negative Symptoms in Schizophrenia
Acronym: NST-SPARK-1b
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Shore Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NST-SPARK-1b
Record Dates: First submitted 2024-01-26; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Negative Symptoms in Schizophrenia; Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Digital Therapeutic; Schizoaffective disorder; Negative Symptoms
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: A group of participants will be introduced to the device and preliminary feasibility, acceptability, and initial target engagement will be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SSD (Experimental): The study design for participants with SSD is a single-arm open-label intervention study. We will collect descriptive information on feasibility and acceptability. Changes in defeatist beliefs and attitudes toward behavioral changes will be evaluated by comparing self-reported ratings before the app intervention vs. immediately afterward and at the 1-week follow-up. All visits will be conducted over video conference with a trained research coordinator.
  Interventions: Device: SPARK

INTERVENTIONS:
Device: SPARK — A gamified augmented reality activity to recapitulate the beginning activation and engagement phase of each recovery-oriented cognitive therapy (CT-R) session

SUMMARY:
This study evaluates the feasibility and acceptability of a prototype for NST-SPARK (version 1.5). This is an augmented reality (AR) mobile phone application that uses Recovery-oriented Cognitive Therapy (CT-R) to target negative symptoms of schizophrenia.

NST-SPARK uses a game AR activity to recapitulate the beginning activation and engagement phase of each CT-R session as per standardized practices for this therapeutic modality.

DETAILED DESCRIPTION:
The specific beliefs targeted during each module are queried before engaging in the AR activity to obtain participant buy in. A self-assessment is taken before and then subsequent prompts challenge these beliefs over the course of the activity. After completion of the AR activity the self-assessment is performed again and the results are compared against the pre-activity responses.

The responses received pre- and then post- activity determine the responses SPARK provides to the participant.

Example: Question: How ambitious or motivated do you feel now?

If the post activity response shows a higher level of motivation compared to the pre-activity assessment the participant will receive the following: So you felt more motivated and more energized! And you did more work not less! Like the more you do the better you feel.

The prototype NST-SPARK v.1.5 has 2 modules: 1) SPARK ENERGY and 2) SPARK MOTIVATION, and is an abbreviated experience following the general framework for NST-SPARK.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-5 criteria for schizophrenia, schizoaffective disorder, schizophreniform disorder, or unspecified psychotic disorder.
* Presence of negative symptoms - SANS rating of 2 or higher on either Avolition/Apathy or Anhedonia/Asociality subscale.
* Capacity to understand the study procedures and provide informed consent.
* Has dependable access to a device with videoconferencing capability and stable wifi connection which can be accessed by the study iPhone.
* Proficient in English.

Exclusion Criteria:

* Recent change in level of care: antipsychotic medication changes in the last 4 weeks OR hospitalization or emergency room/crisis visits in the last 12 weeks.
* Acute safety risk - any indication of ongoing risk to themselves or others.
* Substance induced psychotic disorder or primary mood disorder with psychosis.
* Severe cognitive or physical limitations preventing the participant from being able to independently use NST-SPARK.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of NST-SPARK | This measure will be collected twice: 1) at the first study visit, immediately after using the intervention, and 2) at the 1 week follow-up.
  Measured by average ratings from the self-reported questionnaire (Acceptability of Intervention Measure, scored from 1-5 with 5 representing the highest level of acceptability).
Feasibility of NST-SPARK | This measure will be collected twice: 1) at the first study visit, immediately after using the intervention, and 2) at the 1 week follow-up.
  Measured by average ratings from self-reported questionnaire (Feasibility of Intervention Measure - FIM), scored from 1-5 with 5 representing the highest level of feasibility)
Open-ended feedback about the NST-SPARK user experience | This measure will be collected twice: 1) at the first study visit, immediately after using the intervention, and 2) at the 1 week follow-up.
  Qualitative summary of responses to semi-structured open-ended interview to be conducted with participants, eliciting responses to questions like the following:
  What are your first impressions? What do you like most about the app? What do you like least about the app or what are some areas that need to be improved? Did you experience any negative effects from using the app? For example, dizziness, vertigo, or changes in your symptoms? Do you think you'd be able to use this app from a technical perspective? Does it seem simple enough to operate? If no, which parts seemed confusing or difficult? (Imagine that we added similar but more elaborate experiences for a 12-week long experience, and also provided guides for reaching your goals in the real world.) Would you use this app if your doctor prescribed it for you? What makes you say that?

SECONDARY OUTCOMES:
Changes in defeatist beliefs | This measure will be collected three times: 1) at the first study visit, before using the intervention, 2) at the first study visit, immediately after using the intervention, and 3) at the 1 week follow-up.
  Measured by a self-reported scale (Defeatist Beliefs Scale - 5 items scored from 1-7 with 7 being the lowest level of defeatist beliefs).
Attitude toward goal-oriented activities | This measure will be collected three times: 1) at the first study visit, before using the intervention, 2) at the first study visit, immediately after using the intervention, and 3) at the 1 week follow-up.
  Customized likert scale and semi-structured questions about participant attitudes toward goals they have identified. Results to be reported quantitatively as degree of agreement with statements regarding intention and confidence in making progress toward the goals (scale from 1-5, 5 being the highest level of agreement). Also reporting yes/no and descriptive responses regarding progress toward goals which will be summarized as a percentage of participants who made progress (or not) and as qualitative responses.
Changes in Self Esteem | This measure will be collected three times: 1) at the first study visit, before using the intervention, 2) at the first study visit, immediately after using the intervention, and 3) at the 1 week follow-up.
  Beck Self Esteem Scale with 18 items rated from 1-10 with 10 representing the lowest level of self esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Sunny X Tang, M.D., Principal Investigator — North Shore Therapeutics
Locations (1):
- North Shore Therapeutics, Inc., Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual responses and metadata will be shared for peer review purposes
Supporting Information: Study Protocol, SAP
Time Frame: metadata will become available after study termination for an indefinite period.
Access Criteria: Eligible researchers

REFERENCES:
- [Background] Andreasen NC. The Scale for the Assessment of Negative Symptoms (SANS): conceptual and theoretical foundations. Br J Psychiatry Suppl. 1989 Nov;(7):49-58. No abstract available. PMID 2695141
- [Background] Ascher-Svanum H, Zhu B, Faries DE, Salkever D, Slade EP, Peng X, Conley RR. The cost of relapse and the predictors of relapse in the treatment of schizophrenia. BMC Psychiatry. 2010 Jan 7;10:2. doi: 10.1186/1471-244X-10-2. PMID 20059765
- [Background] Carbon M, Correll CU. Thinking and acting beyond the positive: the role of the cognitive and negative symptoms in schizophrenia. CNS Spectr. 2014 Dec;19 Suppl 1:38-52; quiz 35-7, 53. doi: 10.1017/S1092852914000601. Epub 2014 Nov 18. PMID 25403863
- [Background] Correll CU, Galling B, Pawar A, Krivko A, Bonetto C, Ruggeri M, Craig TJ, Nordentoft M, Srihari VH, Guloksuz S, Hui CLM, Chen EYH, Valencia M, Juarez F, Robinson DG, Schooler NR, Brunette MF, Mueser KT, Rosenheck RA, Marcy P, Addington J, Estroff SE, Robinson J, Penn D, Severe JB, Kane JM. Comparison of Early Intervention Services vs Treatment as Usual for Early-Phase Psychosis: A Systematic Review, Meta-analysis, and Meta-regression. JAMA Psychiatry. 2018 Jun 1;75(6):555-565. doi: 10.1001/jamapsychiatry.2018.0623. PMID 29800949
- [Background] Ford TJ, Buchanan DM, Azeez A, Benrimoh DA, Kaloiani I, Bandeira ID, Hunegnaw S, Lan L, Gholmieh M, Buch V, Williams NR. Taking modern psychiatry into the metaverse: Integrating augmented, virtual, and mixed reality technologies into psychiatric care. Front Digit Health. 2023 Mar 24;5:1146806. doi: 10.3389/fdgth.2023.1146806. eCollection 2023. PMID 37035477
- [Background] Lundin RM, Yeap Y, Menkes DB. Adverse Effects of Virtual and Augmented Reality Interventions in Psychiatry: Systematic Review. JMIR Ment Health. 2023 May 5;10:e43240. doi: 10.2196/43240. PMID 37145841
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459